CLINICAL TRIAL: NCT06202898
Title: Economic Navigation and Strengthening to Research Unrestricted Services for Transgender Women (ENTRUST)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: Sunserve (Unknown); Survivor's Pathway (Unknown); 26Health (Unknown); National Institute of Drug Abuse (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00005488
Record Dates: First submitted 2023-12-21; First posted 2024-01-12 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Transgender Women; Aids; Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — BaseLine dental cement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ENTRUST (Experimental): The proposed intervention 'ENTRUST' will address structural disparities transgender women encounter by providing skills to aid with economic navigation while simultaneously strengthening and improving social cohesion to increase the odds of them linking to care that is available to them.
  Interventions: Other: Baseline; Other: ENTRUST
- Control (Active Comparator): Comparison control group.
  Interventions: Other: Baseline; Other: Control

INTERVENTIONS:
Other: Baseline — At the baseline visits, all study participants will be complete an interviewer-assisted questionnaire using REDCap, and will also receive the SBIRT-T MI-based intervention. Participants randomized to the ENTRUST intervention group will also be assigned to a cohort for strength sessions, and they will be provided with a schedule of strength session visits
Other: ENTRUST — Participants randomized to the ENTRUST intervention group will also be assigned to a cohort for economic strength sessions, group-based economic training through photovoice activities and adapted screening brief intervention and treatment (SBIRT-T) adapted for transgender women delivered by a facilitator or digitally.
  Arms: ENTRUST
Other: Control — participants assigned to the control arm will have the option of participating in the four additional strength sessions.
  Arms: Control

SUMMARY:
The overall hypothesis is that stabilizing transgender women financially while providing them tailored counselling will increase their odds of them linking to substance use services, PrEP services if they do not have HIV, and transgender women who are living with HIV will be more adherent to their ART treatment.

DETAILED DESCRIPTION:
There continues to be a gap in the extant literature on the relationship between substance abuse and achievement of viral suppression (VS) through adherent antiretroviral treatment (ART) or PrEP uptake among transgender women which warrants further investigation. Harmful alcohol and illicit drug use associated with substance use disorders (SUD) have been independently linked to condomless sex and hinder engagement in ending the HIV epidemic (EHE) prevention initiatives, including HIV retention in care and adherence to treatment to achieve viral suppression and PrEP use.

Transgender women are among the most at risk group of sexually active populations, yet least likely to be aware of and/or use preexposure prophylaxis (PrEP) to prevent HIV transmission.5 PrEP and routine HIV/STI screening, are effective approaches to reduce HIV incidence in marginalized at-risk populations and are consistent with the US National HIV/AIDS strategy.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Male at birth
* Identify as a woman/transgender woman
* Should not be consistently using PrEP (less than four doses per week)
* Should not have any known allergy or adverse reaction to PrEP or the active drug tenofovir in ART. One of the goals of the study is to move more people into a PrEP program
* Be able to speak and understand spoken English and/or Spanish (including persons who cannot read or write)
* Have a smart phone that can take pictures

Exclusion Criteria:

* Unwilling to adhere to study procedures
* Participation in an HIV vaccine trial
* Have a life-threatening SUD*
* Any condition, that in the opinion of the study staff, would make participation in the study unsafe, or interfere with achieving the study objective such as medical conditions which prevents the use of PrEP
* Unable to provide consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Identify as a woman/transgender woman
Enrollment: 110 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with substance abuse | 1 year
  The rate of change of substance abuse incidence for both arms

SECONDARY OUTCOMES:
Rate of substance use in transgender women | 1 year
  The rate of stabilizing transgender women financially while providing them tailored counselling to increase their odds of them linking to substance use services, pre-exposure prophylaxis (PrEP) services if they do not have HIV, and transgender women who are living with HIV to be more adherent to their antiretroviral therapy (ART) treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Cyrus, PhD, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States